CLINICAL TRIAL: NCT06863701
Title: Efficacy and Safety Study for the Combination of Etoricoxib / Betamethasone Compared to Etoricoxib for the Treatment of Patients Diagnosed With Acute Gout Arthritis
Brief Title: Efficacy Anda Safety of Etoricoxib With Betamethasone for the Treatment of Acute Gout Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL- 30953 - III - 23 (1)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Gout Arthritis; Gout Attack
Keywords: Gout Arthritis; Gout Attack; Etoricoxib; Betamethasone
MeSH Terms: conditions — Arthritis, Gouty | interventions — Etoricoxib; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib+Betamethasone (Experimental): Administered orally, 1 tablet a day for 8 days.
  Interventions: Drug: Etoricoxib + Betamethasone fixed dose
- Etoricoxib (Active Comparator): Administered orally, 1 pill a day for 8 days.
  Interventions: Drug: Etoricoxib fixed dose

INTERVENTIONS:
Drug: Etoricoxib + Betamethasone fixed dose — One tablet of 90 mg / 0.25 mg a day
  Other Names: Etori + Beta
  Arms: Etoricoxib+Betamethasone
Drug: Etoricoxib fixed dose — One pill of 90 mg a day
  Other Names: Etori
  Arms: Etoricoxib

SUMMARY:
Phase III longitudinal, multicenter, randomized, double-blind clinical trial. The aim of this study is to evaluate the efficacy and safety of the Fixed-Dose Combination of Etoricoxib/Betamethasone Versus Etoricoxib in Patients With Acute Gouty Arthritis

DETAILED DESCRIPTION:
Researchers will compare the fixed-dose combination of Etoricoxib/Betamethasone versus Etoricoxib in acute gouty arthritis by comparing the level of pain in the affected joint during the 8 days of follow up. The adverse events related to the interventions will be registered during follow up.

Participants will:

* Be randomized into one of the 2 intervention groups (A or B)
* Visit the clinic in 3 occasions (day 0, day 5 of follow up and day 8 of follow up)
* In case needed the patient could take 500 mg of acetaminophen, as a rescue medication, previous authorization of de principal investigator

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Women of childbearing potential and sexually active must use an acceptable contraceptive method (barrier and/or hormonal) as determined by the investigator.
* History of hyperuricemia diagnosis (uric acid > 7 mg/dL) reported in medical history or patient interview.
* Clinical diagnosis of acute gouty arthritis with a score of at least 4 based on the following criteria: Male (2 points), history of a similar episode (2 points), symptom onset within the last 24 hours (0.5 points), joint redness (1 point), involvement of the first metatarsophalangeal joint (2.5 points), and hypertension or at least one cardiovascular disease (1.5 points).
* Acute episode characterized by severe pain, inflammation, edema, and erythema in the affected joint (≤ 48 hours before study inclusion).
* In the opinion of the Principal Investigator or treating physician, the patient is eligible for treatment with the investigational product and may benefit clinically

Exclusion Criteria:

* Patients participating in another clinical study involving an investigational treatment or participation in one within the two weeks prior to study initiation.
* Patients whose participation in the study may be influenced (e.g., employment relationship with the research center or sponsor, vulnerable populations, etc.).
* In the investigator's judgment, any condition that affects prognosis and prevents outpatient management, which must be assessed by the principal investigator to determine the patient's eligibility.
* History of severe, progressive, or unstable advanced disease of any kind that may interfere with efficacy and safety evaluations or put the patient at risk.
* Pregnant or breastfeeding patients.
* The study medication is contraindicated for medical reasons.
* History of intolerance or allergic reaction to NSAIDs (nonsteroidal anti-inflammatory drugs), paracetamol, or known hypersensitivity to any component of the formulation.
* Significant history of gastrointestinal disorders (e.g., gastric ulcer, Crohn's disease, ulcerative colitis, gastrointestinal bleeding, etc.).
* History of congestive heart failure (NYHA classification II-IV), established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease (including patients who have recently undergone coronary revascularization or angioplasty).
* Treatment with systemic corticosteroids for the management of acute gouty arthritis within two weeks before study initiation.
* Treatment with NSAIDs within 48 hours prior to study initiation, except for aspirin at cardioprotective doses.
* History of treatment failure with selective COX-2 inhibitors, as reported in medical history or patient interview.
* Presence of acute polyarticular gout affecting more than four joints.
* History of alcohol or drug abuse within the past year.
* Clinical suspicion of joint infection or another joint disease different from acute gouty arthritis.
* History of chronic liver failure (Child-Pugh A, B, and/or C), as reported in medical history or patient interview.
* History of chronic renal failure (glomerular filtration rate <30 ml/min/1.73 m²), as reported in medical history or patient interview.
* Significant history of known coagulation disorders (e.g., Von Willebrand disease, hemophilia, vitamin K deficiency, etc.) or use of anticoagulants, as reported in medical history or patient interview.
* Oncology patients (except for basal cell skin cancer) or patients with severe diseases that, in the investigator's opinion, have a severe prognosis or a life expectancy of less than one year, as well as patients with mental illnesses.
* Patients with symptoms suggestive of active COVID-19 infection (e.g., fever, cough, shortness of breath) and/or contact within the last 14 days with a suspected or confirmed COVID-19 case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Compare the degree of pain in the affected joint (using the Likert pain scale) on days 2, 5, and 8, according to their baseline measurement in each treatment group. | 8 days
  A Likert pain scale is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of four answer statements. The pain should be assessed by the principal investigator or designated physician by asking the patient about the joint experiencing the MOST PAIN at the time of the baseline evaluation and during follow-up.
Number of participants with treatment-related adverse events through the patient's diary record. | 8 days
  To describe the frequency, intensity and causality of the adverse events presented during the clinical trial by treatment group. The adverse events will be registered by the patient in the diary record. Each adverse event will be followed up at the discretion of the researcher.

SECONDARY OUTCOMES:
Compare the degree of inflammation (edema) in the affected joint (using the Likert edema scale) on days 2, 5, and 8 according to the baseline measurement for each treatment group. | 8 days
  A Likert edema scale is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of three answer statements. The evaluation must be conducted by the Site Principal Investigator or designated physician on the most affected joint at baseline and during follow-up.
Compare the degree of inflammation (erythema) in the affected joint (using the Likert edema scale) on days 2, 5, and 8 according to the baseline measurement for each treatment group. | 8 days
  A Likert erythema scale is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of three answer statements. The evaluation must be conducted by the Site Principal Investigator or designated physician on the most affected joint at baseline and during follow-up.
Describe the patient's subjective global assessment of the treatment received at the end of the 8-day follow-up period, by treatment group. | 8 days
  The Investigator must ask the patient the following question:
  "How would you rate the study medication you received for acute gouty arthritis?" at day 8 of follow-up. The assessment would be through a likert scale. The likert scales is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of four answer statements.
Describe the investigator's subjective global assessment of the treatment received by the patient at the end of the 8-day follow-up period, by treatment group. | 8 days
  How would the investigator rate the treatment with the study medication the patient received for acute gouty arthritis?. The question would be assessed through a likert scale. The likert scales is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of four answer statements.

OTHER OUTCOMES:
Report the number of patients who require the use of rescue medication during the clinical trial in each treatment group | 8 days
  The rescue medication will be acetaminophen 500 mg: - The patient that considers the need for rescue medication must call the doctor, who will be in charge of applying the VAS scale by telephone. If the doctor considers it necessary, the taking of the rescue medication will be indicated.
To report the percentage of therapeutic adherence at day 8 of the intervention in each treatment group. | 8 days
  Therapeutic adherence will be defined by the principal researcher. Adherence to treatment will be defined as a consumption ≥ 80% of the doses that the patient should have ingested at the time of the corresponding evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Lanuza-Ramirez, MD, Principal Investigator — Consultorio Médico "Dr. Rodrigo Suárez Otero"; Rodrigo Suarez-Otero, MD, Principal Investigator — SMIQ, S. De. R.L. de C.V. (Grupo Cien y ético de Querétaro)
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li M, Yu C, Zeng X. Comparative efficacy of traditional non-selective NSAIDs and selective cyclo-oxygenase-2 inhibitors in patients with acute gout: a systematic review and meta-analysis. BMJ Open. 2020 Sep 10;10(9):e036748. doi: 10.1136/bmjopen-2019-036748. PMID 32912981
- [Background] van Durme CM, Wechalekar MD, Landewe RB, Pardo Pardo J, Cyril S, van der Heijde D, Buchbinder R. Non-steroidal anti-inflammatory drugs for acute gout. Cochrane Database Syst Rev. 2021 Dec 9;12(12):CD010120. doi: 10.1002/14651858.CD010120.pub3. PMID 34882311
- [Background] Shukla AK, Jhaj R, Misra S, Ahmed SN, Nanda M, Chaudhary D. Agreement between WHO-UMC causality scale and the Naranjo algorithm for causality assessment of adverse drug reactions. J Family Med Prim Care. 2021 Sep;10(9):3303-3308. doi: 10.4103/jfmpc.jfmpc_831_21. Epub 2021 Sep 30. PMID 34760748
- [Background] Man CY, Cheung IT, Cameron PA, Rainer TH. Comparison of oral prednisolone/paracetamol and oral indomethacin/paracetamol combination therapy in the treatment of acute goutlike arthritis: a double-blind, randomized, controlled trial. Ann Emerg Med. 2007 May;49(5):670-7. doi: 10.1016/j.annemergmed.2006.11.014. Epub 2007 Feb 5. PMID 17276548
- [Background] Janssens HJ, Janssen M, van de Lisdonk EH, van Riel PL, van Weel C. Use of oral prednisolone or naproxen for the treatment of gout arthritis: a double-blind, randomised equivalence trial. Lancet. 2008 May 31;371(9627):1854-60. doi: 10.1016/S0140-6736(08)60799-0. PMID 18514729
- [Background] Rainer TH, Cheng CH, Janssens HJ, Man CY, Tam LS, Choi YF, Yau WH, Lee KH, Graham CA. Oral Prednisolone in the Treatment of Acute Gout: A Pragmatic, Multicenter, Double-Blind, Randomized Trial. Ann Intern Med. 2016 Apr 5;164(7):464-71. doi: 10.7326/M14-2070. Epub 2016 Feb 23. PMID 26903390
- [Background] Becker DE. Basic and clinical pharmacology of glucocorticosteroids. Anesth Prog. 2013 Spring;60(1):25-31; quiz 32. doi: 10.2344/0003-3006-60.1.25. PMID 23506281
- [Background] Clarke R, Derry S, Moore RA. Single dose oral etoricoxib for acute postoperative pain in adults. Cochrane Database Syst Rev. 2014 May 8;2014(5):CD004309. doi: 10.1002/14651858.CD004309.pub4. PMID 24809657
- [Background] Xu L, Liu S, Guan M, Xue Y. Comparison of Prednisolone, Etoricoxib, and Indomethacin in Treatment of Acute Gouty Arthritis: An Open-Label, Randomized, Controlled Trial. Med Sci Monit. 2016 Mar 11;22:810-7. doi: 10.12659/msm.895749. PMID 26965791
- [Background] Neilson J, Bonnon A, Dickson A, Roddy E; Guideline Committee. Gout: diagnosis and management-summary of NICE guidance. BMJ. 2022 Aug 30;378:o1754. doi: 10.1136/bmj.o1754. No abstract available. PMID 36041743
- [Background] Pisaniello HL, Fisher MC, Farquhar H, Vargas-Santos AB, Hill CL, Stamp LK, Gaffo AL. Efficacy and safety of gout flare prophylaxis and therapy use in people with chronic kidney disease: a Gout, Hyperuricemia and Crystal-Associated Disease Network (G-CAN)-initiated literature review. Arthritis Res Ther. 2021 Apr 28;23(1):130. doi: 10.1186/s13075-021-02416-y. PMID 33910619
- [Background] Pelaez-Ballestas I, Sanin LH, Moreno-Montoya J, Alvarez-Nemegyei J, Burgos-Vargas R, Garza-Elizondo M, Rodriguez-Amado J, Goycochea-Robles MV, Madariaga M, Zamudio J, Santana N, Cardiel MH; Grupo de Estudio Epidemiologico de Enfermedades Musculo Articulares (GEEMA). Epidemiology of the rheumatic diseases in Mexico. A study of 5 regions based on the COPCORD methodology. J Rheumatol Suppl. 2011 Jan;86:3-8. doi: 10.3899/jrheum.100951. PMID 21196592
- [Background] FitzGerald JD, Dalbeth N, Mikuls T, Brignardello-Petersen R, Guyatt G, Abeles AM, Gelber AC, Harrold LR, Khanna D, King C, Levy G, Libbey C, Mount D, Pillinger MH, Rosenthal A, Singh JA, Sims JE, Smith BJ, Wenger NS, Bae SS, Danve A, Khanna PP, Kim SC, Lenert A, Poon S, Qasim A, Sehra ST, Sharma TSK, Toprover M, Turgunbaev M, Zeng L, Zhang MA, Turner AS, Neogi T. 2020 American College of Rheumatology Guideline for the Management of Gout. Arthritis Rheumatol. 2020 Jun;72(6):879-895. doi: 10.1002/art.41247. Epub 2020 May 11. PMID 32390306